CLINICAL TRIAL: NCT02046213
Title: An Open-label, Single-dose Study to Determine the Metabolism and Excretion of [14C]E2006 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-007
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Metabolism and Excretion
Keywords: Metabolism and Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E2006 (Experimental): Single oral 10mg dose of 100 uCi [14C]E2006
  Interventions: Drug: E2006

INTERVENTIONS:
Drug: E2006 — Single oral 10mg dose of 100 uCi [14C]E2006

SUMMARY:
The purpose of this study is to determine the metabolism and excretion of [14C]E2006 in healthy male subjects.

DETAILED DESCRIPTION:
This is an open-label, single-dose study in healthy male subjects. The study will have 2 phases: Pretreatment and Treatment. The Pretreatment Phase will last up to 21 days and will consist of a Screening Period and a Baseline Period, during which each subject's eligibility will be determined and assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male 18 to 55 years, inclusive, at the time of informed consent
2. Body mass index (BMI) of 18 to 32 kg/m2 at Screening
3. Must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must not be of childbearing potential or must be practicing highly effective contraception throughout the study period and for 90 days after study drug discontinuation. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.
4. Provide written informed consent
5. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

1. Participated in a 14C research study within the 6 months prior to Day -2. The total radiation exposure to radiolabelled compounds from this study and any previous studies must be within the recommended levels considered safe (per US 21 CFR 361.1)
2. Exposure to clinically significant radiation (greater than 100 milliseiverts) within 12 months prior to Day -2
3. Any history of cerebrovascular disease (stroke or transient ischemic attack)
4. A prolonged QT/QTc interval (QTc greater than 450 msec) as demonstrated upon confirmatory ECG if first ECG indicates prolonged QT/QTc interval
5. History of prolonged QT/QTc interval
6. History of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
7. Heart rate less than 40 or greater than 100 beats/min at Screening or Baseline
8. History of ischemic heart disease (e.g., acute coronary syndromes, stable angina), syncope or cardiac arrhythmias
9. Systolic blood pressure greater than 140 mmHg or less than 90 mmHg or diastolic blood pressure greater than 90 mmHg or less than 60 mmHg at Screening or Baseline
10. Hemoglobin less than 12.5 g/dL or hemotocrit less than or equal to 38% at Baseline check-in
11. Evidence of clinically significant disease (e.g., psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system) that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments
12. Any laboratory abnormalities considered clinically significant by the investigator
13. Clinically significant illness which required medical treatment within 8 weeks of dosing or a clinically significant infection within 4 weeks of dosing
14. Any history of gastrointestinal surgery (e.g., hepatectomy, nephrotomy, digestive organ resection) that may affect PK profiles of study drugs
15. Hypersensitivity to the study drug or any of its excipients
16. Known to be human immunodeficiency virus (HIV) positive or positive on viral screen for HIV or viral hepatitis B or hepatitis C
17. History of drug or alcohol dependency or abuse within approximately the last 2 years or who have a positive urine drug test or breath alcohol test at Screening or Baseline
18. Do not meet the restrictions on concomitant medications, food and beverages (see below)
19. Use of illegal (or legalized) recreational drugs in the past year
20. Engagement in strenuous exercise within 2 weeks prior to dosing (e.g., marathon runners, weight lifters)
21. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days preceding informed consent

    Restrictions on prior and concomitant medications, food and beverages
22. Prescription drugs are prohibited within 4 weeks of dosing and over-the-counter drugs within 2 weeks prior to dosing or throughout the Treatment Period
23. Smoking or use of tobacco or nicotine-containing products is prohibited within 4 weeks prior to dosing and throughout the Treatment Period
24. Intake of caffeinated beverages or food is prohibited within 72 hours prior to dosing and until 72 hours postdose
25. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect CYP3A4 enzyme or transporters (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) is prohibited within 2 weeks prior to dosing and throughout the Treatment Period
26. Intake of herbal preparations containing St. John's Wort is prohibited within 4 weeks prior to dosing and throughout the Treatment Period
27. Any subject that has a known history of malaria or has traveled to a country with known malarial risk (ie, designated as a 'high' or 'moderate' risk country according to the list available athttp://www.cdc.gov/malaria) within the last year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Excretion of E2006: urine/feces concentration | Up to 35 days
  Total radioactivity derived from [14C]E2006-related material and E2006 will be analyzed in urine and feces. [14C]E2006 radiolabeled material will be quantified in urine and feces for total radioactivity using a scintillation counting method and/or an accelerator mass spectrometry.
Pharmacokinetics: Plasma concentration of E2006/metabolite | Up to 816 hours postdose
  Total radioactivity derived from [14C]E2006-related material, E2006, and metabolites will be analyzed in whole blood, plasma, and red blood cells. [14C]E2006 radiolabeled material will be quantified in whole blood, plasma, red blood cells for total radioactivity using a scintillation counting method and/or accelerator mass spectrometry.

SECONDARY OUTCOMES:
Pharmacokinetics: Metabolic profile of E2006: plasma/urine/feces concentration | Urine/Feces: Up to 35 days; Plasma: Up to 816 hours postdose
  Metabolite profiling in plasma, urine, and feces will be performed by radio-high performance liquid chromatography (radio-HPLC) methods. Metabolites will be identified on the radiochromatograms, and the amount of the each metabolite will be quantified based on the peak areas on the chromatograms. For metabolites detected on the radiochromatograms, LC/MS/MS analysis will be performed to estimate and identify their chemical structures.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States